CLINICAL TRIAL: NCT03531918
Title: A Single-Center Phase 1/2 Study of Single- or Fractioned-Dose Gemtuzumab Ozogamicin in Combination With G-CSF, Cladribine, Cytarabine, and Mitoxantrone for Previously Untreated Adult Acute Myeloid Leukemia or High-Grade Myeloid Neoplasm
Brief Title: Gemtuzumab Ozogamicin With G-CSF, Cladribine, Cytarabine & Mitoxantrone for Untreated AML & High-Grade Myeloid Neoplasm
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Roland B Walter, Professor, Clinical Research Division, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10000; NCI-2018-00776 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10000 (Other: Fred Hutch/University of Washington Cancer Consortium); RG9218023 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2018-05-09; First posted 2018-05-22 (Actual); Results first posted 2022-11-04 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cladribine; Cytarabine; Gemtuzumab; pegylated granulocyte colony-stimulating factor; Mitoxantrone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (GO, GCLAM) (Experimental): INDUCTION THERAPY: Participants receive gemtuzumab ozogamicin IV either as a single dose on day 1, or as three doses on days 1, 4, and 7. Participants also receive G-CSF SC on days 0-5, cladribine IV over 2 hours on days 1-5, cytarabine IV over 2 hours on days 1-5, and mitoxantrone hydrochloride IV on days 1-3. Patients who do not achieve a CR or CRi following the first cycle of induction are eligible for a second cycle, which is given without gemtuzumab ozogamicin. Participants with a CR or CRi may then proceed to Post-Remission Therapy.
  POST-REMISSION THERAPY: Participants receive G-CSF, cladribine, and cytarabine as in Induction Therapy during cycle 1, and cytarabine IV every 12 hours on days 1-6 of cycles 2-3. Treatment repeats every month for up to 3 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cladribine; Drug: Cytarabine; Drug: Gemtuzumab Ozogamicin; Biological: Recombinant Granulocyte Colony-Stimulating Factor; Other: Laboratory Biomarker Analysis; Drug: Mitoxantrone Hydrochloride

INTERVENTIONS:
Drug: Cladribine — Given IV
  Other Names: 2-CdA; 2CDA; CdA; Cladribina; Leustat; Leustatin; Leustatine; RWJ-26251
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Gemtuzumab Ozogamicin — Given IV
  Other Names: Calicheamicin-Conjugated Humanized Anti-CD33 Monoclonal Antibody; CDP-771; CMA-676; gemtuzumab; hP67.6-Calicheamicin; Mylotarg; WAY-CMA-676
Biological: Recombinant Granulocyte Colony-Stimulating Factor — Given SC
  Other Names: 143011-72-7; Recombinant Colony-Stimulating Factor 3; rhG-CSF
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mitoxantrone Hydrochloride — Given IV
  Other Names: CL 232315; DHAD; DHAQ; Dihydroxyanthracenedione Dihydrochloride; Mitoxantrone Dihydrochloride; Mitoxantroni Hydrochloridum; Mitozantrone Hydrochloride; Mitroxone; Neotalem; Novantrone; Onkotrone; Pralifan

SUMMARY:
This phase I/II trial studies the side effects and best dosing frequency of gemtuzumab ozogamicin when given in combination with granulocyte colony stimulating factor (G-CSF), cladribine, cytarabine and mitoxantrone (GCLAM) and to see how well they work in treating participants with acute myeloid leukemia or high-grade myeloid tumors (neoplasms) that have not been previously treated. Antibody-drug conjugates, such as gemtuzumab ozogamicin, act by directly delivering toxic chemotherapy to cancer cells. Granulocyte colony stimulating factor is a growth factor used to stimulate leukemia cells and render them more sensitive to chemotherapy drugs. Drugs used in chemotherapy, such as cladribine, cytarabine and mitoxantrone, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving gemtuzumab ozogamicin in combination with G-CSF, cladribine, cytarabine and mitoxantrone hydrochloride may work better in treating participants with acute myeloid leukemia or high-grade myeloid neoplasm.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum-tolerated dose (MTD) of gemtuzumab ozogamicin (GO) when added to GCLAM in patients with newly-diagnosed AML requiring induction chemotherapy. (Phase I) II. To evaluate the 6-month and 1-year event-free survival (EFS) rate with GO + GCLAM treated at the MTD. (Phase II)

SECONDARY OBJECTIVES:

I. Describe, within the limits of a phase 1/2 study, the toxicity profile of the study regimen.

II. Compare, within the limits of a phase 1/2 study, measurable residual disease (MRD) rates with GO + GCLAM at the MTD to patients treated previously with GCLAM alone.

III. Estimate, within the limits of a phase 1/2 study, the relationship between MRD status after induction therapy and relapse risk/time to relapse as well as relapse-free and overall survival.

IV. Compare, within the limits of a phase 1/2 study, complete remission rates with GO + GCLAM at the MTD to patients treated previously with GCLAM alone.

V. Compare, within the limits of a phase 1/2 study, overall survival rates with GO + GCLAM at the MTD to patients treated previously with GCLAM alone VI. Evaluate, within the limits of a phase 1/2 study, the impact of GO dosing regimens on the duration of cytopenias.

VII. Collect biological specimens for use for the future laboratory investigation of biomarkers for response to GO.

OUTLINE: This is a phase I dose escalation study of gemtuzumab ozogamicin followed by a phase II study.

INDUCTION THERAPY: Participants receive gemtuzumab ozogamicin intravenously (IV) either as a single dose on day 1, or as three doses on days 1, 4, and 7. Participants also receive G-CSF subcutaneously (SC) on days 0-5, cladribine IV over 2 hours on days 1-5, cytarabine IV over 2 hours on days 1-5, and mitoxantrone hydrochloride IV on days 1-3. Patients who do not achieve a CR or CRi following the first cycle of induction are eligible for a second cycle, which is given without gemtuzumab ozogamicin. Participants with a complete remission (CR) or complete remission with incomplete count recovery (CRi) may then proceed to Post-Remission Therapy.

POST-REMISSION THERAPY: Participants receive G-CSF, cladribine, and cytarabine as in Induction Therapy during cycle 1, and cytarabine IV every 12 hours on days 1-6 of cycles 2-3. Treatment repeats every month for up to 3 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up every 3 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of untreated "high-grade" myeloid neoplasm (≥ 10% blasts in blood or bone marrow) or acute myeloid leukemia (AML) other than acute promyelocytic leukemia (APL) with t(15;17)(q22;q12) or variants according to the 2016 World Health Organization (WHO) classification; outside diagnostic material is acceptable to establish diagnosis; submission of peripheral blood specimen for flow cytometry performed at the study institution should be considered; diagnostic material must have been submitted for cytogenetic and/or molecular testing as clinically appropriate
* Medically fit, as defined by treatment-related mortality (TRM) score ≤13.1 calculated with simplified model
* The use of hydroxyurea prior to study registration is allowed; patients with symptoms/signs of hyperleukocytosis or white blood cells (WBC) > 100,000/uL can be treated with leukapheresis or may receive up to 2 doses of cytarabine (up to 500 mg/m^2/dose) prior to enrollment
* Patients may have received low-intensity treatment (e.g. azacitidine/decitabine, lenalidomide, growth factors) for antecedent low-grade myeloid neoplasm (i.e. < 10% blasts in blood and bone marrow)
* Bilirubin ≤ 2.5 x institutional upper limit of normal (IULN) unless elevation is thought to be due to hepatic infiltration by AML, Gilbert's syndrome, or hemolysis (assessed within 14 days prior to study day 0)
* Serum creatinine ≤ 2.0 mg/dL (assessed within 14 days prior to study day 0)
* Left ventricular ejection fraction ≥ 45%, assessed within 12 months prior to study day 0, e.g. by multigated acquisition (MUGA) scan or echocardiography, or other appropriate diagnostic modality and no clinical evidence of congestive heart failure
* Women of childbearing potential and men must agree to use adequate contraception
* Provide written informed consent

Exclusion Criteria:

* Myeloid blast crisis of chronic myeloid leukemia (CML), unless patient is not considered candidate for tyrosine kinase inhibitor treatment
* Concomitant illness associated with a likely survival of < 1 year
* Active systemic fungal, bacterial, viral, or other infection, unless disease is under treatment with anti-microbials, and/or controlled or stable (e.g. if specific, effective therapy is not available/feasible or desired [e.g. known chronic viral hepatitis, human immunodeficiency virus (HIV)]); patient needs to be clinically stable as defined as being afebrile and hemodynamically stable for 24 hours; patients with fever thought to be likely secondary to leukemia are eligible
* Known hypersensitivity to any study drug
* Confirmed or suspected pregnancy or active breast feeding
* Treatment with any other investigational anti-leukemia agent; in phase 2, treatment with a tyrosine kinase inhibitor for patients with FLT3-mutated AML is permissible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roland Walter, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- GO1 Dose Level Phase 1: Participants received 1 dose of gemtuzumab ozogamicin (GO) intravenously at 3 mg/m2 per dose on day 1.
  All doses of GO were capped at 4.5 mg.
- GO3 Dose Level Includes Phase 1 and Phase 2: Phase 1: Participants received 3 doses of gemtuzumab ozogamicin (GO) intravenously at 3 mg/m2 per dose on days 1, 4, and 7.
  Phase 2: Participants received CLAG-M(cladribine, high-dose cytarabine, G-CSF and dose-escalated mitoxantrone)/GO at the recommended phase 2 dose (RP2D) identified in phase 1.
  All doses of GO were capped at 4.5 mg.
Period: Overall Study
Arm/Group | GO1 Dose Level Phase 1 | GO3 Dose Level Includes Phase 1 and Phase 2
Started | 6 | 60
Completed | 6 | 56
Not Completed | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GO1 Dose Level Phase 1 | GO3 Dose Level Includes Phase 1 and Phase 2 | Total
Number analyzed (Participants) | 6 | 60 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 28 | 30
  >=65 years | 4 | 32 | 36
Age, Continuous [Median (Full Range); unit: years] | 64.83 [51 to 73] | 61.13 [19 to 80] | 61.47 [19 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 28 | 32
  Male | 2 | 32 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 5 | 45 | 50
  Unknown or Not Reported | 0 | 12 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 1 | 1
  White | 5 | 42 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 11 | 11
Region of Enrollment [Number; unit: participants]
  United States | 6 | 60 | 66

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Gemtuzumab Ozogamicin (GO) When Added to GCLAM (Phase 1)
Description: Defined as the highest dose studied in which the incidence of Dose Limiting Toxicity (DLT) is ≤33% (≤4 of 12 patients experiencing DLT), defined as any Grade 3 non-hematologic toxicity lasting >48 hours that results in >7-day delay of the subsequent treatment cycle, with the exception of febrile neutropenia or infection or toxicities secondary to febrile neutropenia or infection, or any Grade ≥4 non-hematologic toxicity except febrile neutropenia/infection (or toxicities secondary to febrile neutropenia or infection) unless felt to be a direct consequence of treatment-related toxicity (e.g. intestinal infection following mucosal barrier breakdown), and with the exception of constitutional symptoms if recovery to Grade ≤2 within 14 days. The National Cancer Institute Common Terminology Criteria for Adverse Events v5.0 will be used.
Time Frame: At time of count recovery, second cycle of treatment, response assessment or removal from protocol (at approximately 1 month).
Measure: Count of Participants; unit: Participants
Arm/Group | GO1 Dose Level Phase 1 | GO3 Dose Level Includes Phase 1 and Phase 2
Number analyzed (Participants) | 6 | 60
Participants | NA — The Maximum Tolerated Dose was not reached since the GO3 dose level (the maximum dose specified by the protocol) had a dose-limiting toxicity rate of greater than 33%. Thusly, the GO3 dose level is the recommended phase 2 dose but not the MTD. | NA — The Maximum Tolerated Dose was not reached since the GO3 dose level (the maximum dose specified by the protocol) had a dose-limiting toxicity rate of greater than 33%. Thusly, the GO3 dose level is the recommended phase 2 dose but not the MTD.

2. Primary Outcome: Event-free Survival (EFS) Rate (Phase 2)
Description: A two-stage design will be used to evaluate the EFS. Patients treated at the maximum tolerated dose (MTD) from the phase 1 portion of the trial will be used in the phase 2 analysis. If censoring occurs, secondary analyses analyzing 6-month or 1-year EFS accounting for censoring will be done, including estimating 6-month or 1-year EFS using the Kaplan-Meier method. The first stage of the two-stage phase 2 design will evaluate 30 patients. If 20 or more of the first 30 patients are alive without event at 6-months after study registration, an additional 30 patients will be enrolled. If 46 or more of the 60 patients treated at the MTD are alive and without event at 6-months after study registration, the study will consider the regimen of interest for further investigation. Patients last known to be alive in CR were censored at date of last contact.
Time Frame: From the start of study treatment, assessed at 6 months and 1 year
Population: GO1 participants were treated in dose escalation. The primary endpoint per protocol is to assess the EFS rate at the MTD or RP2D and was not assessed at dose levels below the RP2D.
Measure: Number (95% Confidence Interval); unit: percent of participants
Groups:
- GO1 Dose Level: Participants received 1 dose of gemtuzumab ozogamicin (GO) intravenously at 3 mg/m2 per dose on day 1.
  All doses of GO were capped at 4.5 mg.
Arm/Group | GO1 Dose Level | GO3 Dose Level Includes Phase 1 and Phase 2
Number analyzed (Participants) | 0 | 60
percent of participants
  Event-free Survival (6 months) |  | 73 [63 to 85]
  Event-free survival (12 months) |  | 58 [47 to 72]

3. Secondary Outcome: 30-day All-cause Mortality
Description: As a summary of adverse events (captured on trial using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0), 30-day all cause mortality is reported as a percent of patients treated at the MTD/RP2D.
  Will be estimated and 95% confidence intervals will be calculated. Regression models (logistic regression for binary endpoints, Cox regression for time-to-event endpoints [Cox models for the hazard of the subdistribution for events with competing risks]) will be used to compare outcomes with patients who have received GCLAM without GO at our institution, controlling for measured prognostic factors.
Time Frame: Up to 5 years. 30-day all-cause mortality is reported
Population: 30-day mortality is reported among patients treated at the MTD/RP2D. There is no study-related reason to report survival data on the GO1 dose level. No efficacy assessments were evaluated during the GO1 phase 1 dose escalation study which focuses on DLT/toxicity assessments.
Measure: Number (95% Confidence Interval); unit: proportion died on/before day 30
Arm/Group | GO1 Dose Level Phase 1 | GO3 Dose Level Includes Phase 1 and Phase 2
Number analyzed (Participants) | 0 | 60
proportion died on/before day 30 |  | .03 [.0004 to .12]

4. Secondary Outcome: Relapse-free Survival of GO3 Cohort
Description: RFS was calculated for participants who achieved a complete remission (with or without count recovery; CR or CRi) and measured from the date remission to the first of relapse from CR/CRi or death from any cause. Patients last known to be alive in CR /CRi were censored at date of last contact. Will be estimated using the Kaplan-Meier method. Time to relapse will be estimated using non-parametric estimates of the cumulative incidence curve with death analyzed as a competing event. Regression models (logistic regression for binary endpoints, Cox regression for time-to-event endpoints [Cox models for the hazard of the subdistribution for events with competing risks]) will be used to compare outcomes with patients who have received GCLAM without GO at our institution, controlling for measured prognostic factors.
Time Frame: Up to 5 years. 2-year RFS reported.
Population: RFS is reported among patients treated at the MTD/RP2D. There is no study-related reason to report survival data on the GO1 dose level. No efficacy assessments were evaluated during the GO 1 phase 1 dose escalation study which focuses on DLT/toxicity assessments.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GO1 Dose Level Phase 1 | GO3 Dose Level Includes Phase 1 and Phase 2
Number analyzed (Participants) | 0 | 52
percentage of participants |  | 51 [34 to 64]

5. Secondary Outcome: Overall Survival
Description: OS was calculated for all participants and measured from initial trial therapy to death from any cause. Patients last known ot be alive were censored at date of last contact. Will be estimated using the Kaplan-Meier method. Regression models (logistic regression for binary endpoints, Cox regression for time-to-event endpoints [Cox models for the hazard of the subdistribution for events with competing risks]) will be used to compare outcomes with patients who have received GCLAM without GO at our institution, controlling for measured prognostic factors.
Time Frame: 3 years and 1 month
Population: RFS is reported among patients treated at the MTD/RP2D. There is no study-related reason to report survival data on the GO1 dose level. No efficacy assessments were evaluated during the GO1 phase 1 dose escalation study which focuses on DLT/toxicity assessments.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- GO3 Dose Level: Phase 1: Participants received 3 doses of gemtuzumab ozogamicin (GO) intravenously at 3 mg/m2 per dose on days 1, 4, and 7.
  Phase 2: Participants received CLAG-M(cladribine, high-dose cytarabine, G-CSF and dose-escalated mitoxantrone)/GO at the recommended phase 2 dose (RP2D) identified in phase 1.
  All doses of GO were capped at 4.5 mg.
Arm/Group | GO1 Dose Level Phase 1 | GO3 Dose Level
Number analyzed (Participants) | 0 | 60
percentage of participants |  | 60 [48 to 73]

6. Secondary Outcome: Measurable Residual Disease (MRD) Rates and Remission Rates: CR
Description: Will be estimated and 95% confidence intervals will be calculated. Regression models (logistic regression for binary endpoints, Cox regression for time-to-event endpoints [Cox models for the hazard of the subdistribution for events with competing risks]) will be used to compare outcomes with patients who have received GCLAM without GO at our institution, controlling for measured prognostic factors.
  Complete response (CR) rate is defined as the frequency of patients achieving CR, which is defined by the European LeukemiaNet 2017 guidelines as bone marrow blasts <5%; absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; ANC ≥1.0 x 109/L (1000/mL); platelet count ≥100 x 109/L. (100 000/mL). MRD negative (MRDneg) status is defined as negative for leukemic markers by multiparameter flow cytometry.
  Aplasia was defined as absence of tumoral cells but cellularity not meeting criteria for MLFS.
  Statistical significance tests were not performed.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | GO1 Dose Level Phase 1 | GO3 Dose Level Includes Phase 1 and Phase 2
Number analyzed (Participants) | 6 | 60
Participants
  MRDneg | 4 | 38
  MRDpos | 0 | 7

7. Secondary Outcome: Measurable Residual Disease (MRD) and Remission Rates: CRi (MRDneg)
Description: Will be estimated and 95% confidence intervals will be calculated. Regression models (logistic regression for binary endpoints, Cox regression for time-to-event endpoints [Cox models for the hazard of the subdistribution for events with competing risks]) will be used to compare outcomes with patients who have received GCLAM without GO at our institution, controlling for measured prognostic factors.
  Complete response with incomplete hematologic recovery (CRi) rate is defined as the frequency of patients achieving CRi, which is defined by the European LeukemiaNet 2017 guidelines as all CR criteria except for residual neutropenia (ANC <1.0 x 109/L [1000/mL]) or thrombocytopenia (platelet count <100 x 109/L [100,000/mL]). MRD negative (MRDneg) status is defined as negative for leukemic markers by multiparameter flow cytometry.
  Aplasia was defined as absence of tumoral cells but cellularity not meeting criteria for MLFS.
  Statistical significance tests were not performed.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | GO1 Dose Level Phase 1 | GO3 Dose Level Includes Phase 1 and Phase 2
Number analyzed (Participants) | 6 | 60
Participants | 1 | 7

8. Secondary Outcome: Measurable Residual Disease (MRD) and Remission Rates: CR/CRi
Description: Will be estimated and 95% confidence intervals will be calculated. Regression models (logistic regression for binary endpoints, Cox regression for time-to-event endpoints [Cox models for the hazard of the subdistribution for events with competing risks]) will be used to compare outcomes with patients who have received GCLAM without GO at our institution, controlling for measured prognostic factors.
  Complete response (CR) + complete response with incomplete hematologic recovery (CRi) rate is defined as the frequency of patients achieving CR or CRi per the European LeukemiaNet 2017 criteria as defined above. MRD negative (MRDneg) status is defined as negative for leukemic markers by multiparameter flow cytometry.
  Aplasia was defined as absence of tumoral cells but cellularity not meeting criteria for MLFS.
  Statistical significance tests were not performed.
Time Frame: 90 days
Population: GO1: remission rates for 6 patients: CR rate was 4/6, CR+CRi rate was 5/6 (all MRDneg)
Measure: Count of Participants; unit: Participants
Arm/Group | GO1 Dose Level Phase 1 | GO3 Dose Level Includes Phase 1 and Phase 2
Number analyzed (Participants) | 6 | 60
Participants | 5 | 52

9. Secondary Outcome: Measurable Residual Disease (MRD) and Remission Rates: MLFS (MRDneg)
Description: Will be estimated and 95% confidence intervals will be calculated. Regression models (logistic regression for binary endpoints, Cox regression for time-to-event endpoints [Cox models for the hazard of the subdistribution for events with competing risks]) will be used to compare outcomes with patients who have received GCLAM without GO at our institution, controlling for measured prognostic factors.
  Morphologic leukemia free state (MLFS) rate is defined as the frequency of patients achieving MLFS, which is defined by the European LeukemiaNet guidelines as bone marrow blasts <5%; absence of blasts with Auer rods; absence of extramedullary disease; no hematologic recovery required. At least 200 cells should be enumerated or cellularity should be at least 10%. MRD negative (MRDneg) status is defined as negative for leukemic markers by multiparameter flow cytometry.
  Aplasia was defined as absence of tumoral cells but cellularity not meeting criteria for MLFS.
  Statistical significance
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | GO1 Dose Level Phase 1 | GO3 Dose Level Includes Phase 1 and Phase 2
Number analyzed (Participants) | 6 | 60
Participants | 0 | 2

10. Secondary Outcome: Measurable Residual Disease (MRD) and Remission Rates: Alapasia (MRDneg)
Description: Will be estimated and 95% confidence intervals will be calculated. Regression models (logistic regression for binary endpoints, Cox regression for time-to-event endpoints [Cox models for the hazard of the subdistribution for events with competing risks]) will be used to compare outcomes with patients who have received GCLAM without GO at our institution, controlling for measured prognostic factors.
  o Aplasia rate is defined in this protocol as frequency of patients without blood count recovery after chemotherapy and bone marrow examination showing hypocellularity not meeting cellularity criteria for morphologic leukemia free state (MLFS). MRD negative (MRDneg) status is defined as negative for leukemic markers by multiparameter flow cytometry.
  Aplasia was defined as absence of tumoral cells but cellularity not meeting criteria for MLFS.
  Statistical significance tests were not performed.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | GO1 Dose Level Phase 1 | GO3 Dose Level Includes Phase 1 and Phase 2
Number analyzed (Participants) | 6 | 60
Participants | 0 | 2

ADVERSE EVENTS:
Time Frame: Serious adverse events and other (not including serious) adverse events were monitored and recorded for only the first cycle of therapy (the only period of experimental therapy). Patients were monitored from the start of the first drug administration (on day 0 or day 1) until the start of the second cycle of therapy, or until 1 month post the first response assessment. All-Cause Mortality was assessed for 3 years and 1 month.
Description: Adverse events were collected systematically through regular investigator and study staff assessment in combination with reviews of clinical, laboratory, and imaging records and ongoing direct communication with treating physicians and sub-investigators. Only adverse events rated grade 3 or higher, with the exception of all hematologic toxicities, are recorded, graded, and reported. Grading drawn from CTCAE version 5.0.
Arm/Group | GO1 Dose Level Phase 1 | GO3 Dose Level Includes Phase 1 and Phase 2
All-Cause Mortality (participants affected / at risk) | 0/6 | 2/60
Serious Adverse Events (participants affected / at risk) | 1/6 | 10/60
Other Adverse Events (participants affected / at risk) | 6/6 | 59/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GO1 Dose Level Phase 1 (N=6) | GO3 Dose Level Includes Phase 1 and Phase 2 (N=60)
Grade 4 Bronchopulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Grade 3 Left Ventricular Systolic Dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Grade 4 Aspartate Aminotransferase Increase (Investigations) | 0 (0) | 1 (1)
Grade 3 Reversible Posterior Leukoencephalopathy Syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Grade 3 Intercranial Hemorrhage (Nervous system disorders) | 0 (0) | 2 (2)
Grade 3 Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Grade 4 Tumor Lysis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Grade 3 Pericardial Effusion (Cardiac disorders) | 0 (0) | 1 (1)
Grade 3 Hip Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Grade 4 Upper Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Grade 3 Encephalitis Infection (Infections and infestations) | 0 (0) | 1 (1)
Grade 3 Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Grade 4 Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Grade 4 Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Grade 4 Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GO1 Dose Level Phase 1 (N=6) | GO3 Dose Level Includes Phase 1 and Phase 2 (N=60)
Grade 3 Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 56 (88)
Grade 3 Esophageal Hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Grade 3 Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Grade 3 Enterocolitis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Grade 3 Chest Pain - Cardiac (Cardiac disorders) | 1 (1) | 0 (0)
Grade 3 Sepsis (Infections and infestations) | 2 (2) | 28 (28)
Grade 4 Sepsis (Infections and infestations) | 0 (0) | 3 (4)
Grade 3 Hypotension (Cardiac disorders) | 1 (1) | 1 (2)
Grade 3 Hypertension (Vascular disorders) | 1 (2) | 37 (79)
Grade 3 Skin Infection (Infections and infestations) | 1 (1) | 3 (3)
Grade 3 Headache (Nervous system disorders) | 1 (1) | 0 (0)
Grade 3 Lung Infection (Infections and infestations) | 1 (1) | 7 (9)
Grade 3 Perineal Pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Grade 3 Vaginal Hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Grade 3 Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Grade 3 Alanine Aminotransferase Increase (Investigations) | 0 (0) | 2 (2)
Grade 3 Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Grade 4 Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Grade 3 Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Grade 3 Upper Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 (0) | 4 (4)
Grade 3 Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3)
Grade 3 Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Grade 3 Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 0 (0) | 5 (5)
Grade 3 Urinary Tract Infection (Infections and infestations) | 0 (0) | 2 (2)
Grade 3 Intracranial Hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Grade 3 Aspartate Aminotransferase Increase (Investigations) | 0 (0) | 4 (4)
Grade 3 Hepatic Infection (Infections and infestations) | 0 (0) | 1 (1)
Grade 3 Typhlitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Grade 3 Left Ventricular Systolic Dysfunction (Cardiac disorders) | 0 (0) | 5 (5)
Grade 3 Ejection Fraction Decrease (Investigations) | 0 (0) | 1 (1)
Grade 3 Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Grade 3 Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (7)
Grade 3 Atrial Fibrillation (Cardiac disorders) | 0 (0) | 3 (4)
Grade 3 Myocardial Infarction (Cardiac disorders) | 0 (0) | 2 (2)
Grade 3 Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Grade 4 Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Grade 3 Hematuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Grade 3 Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 6 (6)
Grade 3 Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Grade 3 Esophagitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Grade 3 Mucositis Oral (Gastrointestinal disorders) | 0 (0) | 3 (3)
Grade 3 Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Grade 3 Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Grade 4 Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Grade 3 Hyperphosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Grade 3 Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Grade 3 Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Grade 3 Heart Failure (Cardiac disorders) | 0 (0) | 1 (1)
Grade 3 Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Grade 3 Generalized Edema (General disorders) | 0 (0) | 1 (1)
Grade 3 Catheter Related Infection (Infections and infestations) | 0 (0) | 3 (3)
Grade 3 Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Grade 3 Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Grade 3 Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Grade 3 Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Grade 3 Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Grade 4 Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Grade 3 Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Grade 3 Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Grade 3 Shingles (Infections and infestations) | 0 (0) | 1 (1)
Grade 3 Bronchopulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Grade 3 Dental Caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Grade 3 Colonic Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Grade 3 Colonic Hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Grade 3 Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Grade 3 Anorectal Infection (Infections and infestations) | 0 (0) | 1 (1)
Grade 3 Menorrhagia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Grade 3 Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This is a single center study and generalizability to other centers is unclear. This is a non-randomized, single arm study without a contemporaneously enrolled control arm. The number of participants at the phase 1 dose level GO1 was insufficient to perform statistically reliable analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-17): https://cdn.clinicaltrials.gov/large-docs/18/NCT03531918/Prot_SAP_002.pdf
  • Informed Consent Form (2019-04-10): https://cdn.clinicaltrials.gov/large-docs/18/NCT03531918/ICF_003.pdf